CLINICAL TRIAL: NCT04298606
Title: A Phase 0 Study of CIMAvax-EGF Vaccine in Patients Who Are at High Risk for Lung Cancer and Lung Cancer Survivors at Risk for Recurrence
Brief Title: A Vaccine (CIMAvax-EGF) for the Prevention of Lung Cancer Development or Recurrence
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: I 511919; NCI-2019-08720 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 511919 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2020-03-04; First posted 2020-03-06 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Chronic Obstructive Pulmonary Disease; Lung Non-Small Cell Carcinoma; Pneumonia; Stage IB Lung Cancer AJCC v8; Stage II Lung Cancer AJCC v8; Stage IIA Lung Cancer AJCC v8; Stage IIB Lung Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Carcinoma, Non-Small-Cell Lung; Pneumonia; Lung Neoplasms | interventions — CIMAvax EGF

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Prevention (recombinant human EGF-rP64K/montanide ISA 51) (Experimental): LOADING PHASE: Patients receive recombinant human EGF-rP64K/montanide ISA 51 vaccine IM at 0, 2, 4 and 6 weeks in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE PHASE: Patients receive recombinant human EGF-rP64K/montanide ISA 51 vaccine IM Q4W in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Biological: Recombinant Human EGF-rP64K/Montanide ISA 51 Vaccine

INTERVENTIONS:
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Biological: Recombinant Human EGF-rP64K/Montanide ISA 51 Vaccine — Given IM
  Other Names: Center of Molecular Immunology (CIMA) Epidermal Growth Factor (EGF) Vaccine; Center of Molecular Immunology Epidermal Growth Factor Vaccine; CimaVax; CIMAvax EGF; CIMAvax Epidermal Growth Factor Vaccine; CimaVax Vaccine; CIMAvax-EGF; Recombinant Human EGF-P64K/Montanide Vaccine

SUMMARY:
This early phase I trial studies the side effects of a vaccine called CIMAvax-EGF and to see how well it works in preventing lung cancer from developing in patients at high risk for lung cancer or coming back (recurrence) in stage IB-IIIA non-small cell lung cancer survivors. In many cancers such as lung cancer, there is a protein receptor called EGFR (epidermal growth factor receptor) that is overexpressed within these cancers. Activation of EGFR has shown to lead to tumor growth and development. Previous studies have indicated that EGFR activation is present in the airways of cancer-free subjects as well. CIMAvax-EGF vaccine works by causing the body to make antibodies against EGF that is being produced that could be possibly driving the risk for developing cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the efficacy of the vaccine based on circulating EGF and anti-EGF antibodies.

II. To access the molecular profile of blood, bronchial and nasal brushes, and bronchial biopsies to identify molecular markers associated with treatment and response.

III. To establish the safety of recombinant human EGF-rP64K/montanide ISA 51 vaccine (CIMAvax-EGF) treatment in cancer-free individuals using the Cancer Therapy Evaluation Program (CTEP) National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE version 5).

SECONDARY OBJECTIVE:

I. To evaluate quality of life score changes using European Organization for the Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-Core 30 (C30) in patients who are at high risk for development of lung cancer or recurrence during CIMAvax-EGF treatment.

OUTLINE:

LOADING PHASE: Patients receive recombinant human EGF-rP64K/montanide ISA 51 vaccine intramuscularly (IM) at 0, 2, 4 and 6 weeks in the absence of disease progression or unacceptable toxicity.

MAINTENANCE PHASE: Patients receive recombinant human EGF-rP64K/montanide ISA 51 vaccine IM once every 4 weeks (Q4W) in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 60 days.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed no evidence of cancer on computed tomography (CT) scan within 6 months prior to starting treatment
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Patients must have platelets >= 100 x 10^9/L
* Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry

  * Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure
* PATIENTS AT HIGH-RISK FOR LUNG CANCER COHORT ONLY (COHORT A)
* Must have documented at least one risk factor for lung cancer which includes:

  * Moderate to severe chronic obstructive pulmonary disease (COPD) defined as FEV1/FVC ratio <=75%
  * Positive family history of lung cancer defined as a first degree relative
  * Low body mass index (BMI)
  * History of pneumonia within the last 5 years prior to enrollment
  * Occupational exposure such as asbestos, radon and any other that investigator would deem high risk
* Must have quit smoking =< 15 years ago or be a current smoker
* Must have at least 30 pack year smoking history
* Must have documented pulmonary function test within the last 3 years prior to enrollment. If a patient cannot tolerate a pulmonary function test, an incentive spirometry will be acceptable in place of a pulmonary function test
* LUNG CANCER SURVIVOR COHORT ONLY (COHORT B)
* 1. If patient received surgery or any adjuvant therapy for initial diagnosis of lung cancer, it must have been completed at least 3 months prior to enrollment. Prior surgery or any therapy is not required for eligibility
* Confirmed non-small cell lung cancer (NSCLC) stage IA through 3A at initial diagnosis

Exclusion Criteria:

* Clinically inappropriate to have a bronchoscopy procedure
* Known uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, history of clinically significant cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or nursing female participants
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to receive study drug
* Received an investigational agent within 30 days prior to enrollment
* Has known immunosuppressive disease (e.g. human immunodeficiency virus [HIV], acquired immunodeficiency syndrome [AIDS] or other immune depressing disease). Testing is not mandatory
* Patient has known hypersensitivity to the components of the study drugs or any analogs
* History of autoimmune disorder, with exception of patients with vitiligo or endocrine-related autoimmune conditions receiving appropriate hormonal supplementation who are eligible. Systemic use of immunosuppressant drugs such as steroids (except as hormone replacement therapy or short-course supportive medication such as chemotherapy or drug allergy, etc.), azathioprine, tacrolimus, cyclosporine, etc. within 4 weeks before recruitment
* The following special populations are excluded from this study:

  * Cognitively impaired adults/adults with impaired decision-making capacity
  * Individuals who are not yet adults (infants, children, teenagers)
  * Prisoners
  * Pregnant women

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-11-22 (Actual); Primary Completion 2029-11-22 (Estimated); Study Completion 2029-11-22 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with antibody titers >= 1:4000 in response to vaccination | Up to 60 days post treatment
  The response to the vaccine will be measured using circulating EGF and anti-EGF antibodies replicating the results from the Cuban and Roswell trials. Human EGF will be determined by the Roswell Park Flow and Image Cytometry CCSG supported Resource using a commercial enzyme-linked immunosorbent assay (ELISA) assay (R&D Systems, Minneapolis, MN). EGF antibodies will also be determined, by the Roswell Park Flow and Image Cytometry Resource using an in-house assay developed in cooperation with the Centro de Immunologia Molecular in La Habana, Cuba.
Molecular biomarker analysis | Up to 60 days post treatment
  Will access the molecular profile of blood, bronchial brushes, and bronchial biopsies to identify molecular markers associated with treatment and response. Biomarker scores will be analyzed for the molecular profile endpoint to test if they are significantly different post-treatment compared to pre-treatment (via paired t-test) or if a change in biomarker score (post-versus pre-) is significantly different among responders versus nonresponders (via t-test) as defined by histology and circulating levels of EGF ligand and anti-EGF antibodies. In addition to these biomarkers, gene expression signatures will be analyzed. These include gene expression signatures associated with EGFR activity, the high-grade lesion molecular subtype, and the immune-associated signature predictive of progressive/stable lesions compared with regressive lesions.
Number of patients with grade 3, 4 or 5 toxicities that are attributable to recombinant human EGF-rP64K/montanide ISA 51 vaccine (CIMAvax) | Up to 60 days post treatment
  Measured according to Cancer Therapy Evaluation Program (CTEP) National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5. The plausible range for the true (unobserved) event rate will be estimated by the upper one-sided, 95% Jeffrey's interval.

SECONDARY OUTCOMES:
Change in quality of life scores | Baseline up to 12 months
  Will be assessed using European Organization for the Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-Core 30 (C30).

CONTACTS AND LOCATIONS:
Overall Officials: Mary Reid, PhD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States